CLINICAL TRIAL: NCT05758155
Title: The Effect of Creative Drama Education Applied to Nursing Students on Mental Health Literacy Levels: A Randomized Controlled Study
Brief Title: The Effect of Creative Drama on the Level of Mental Health Literacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AİBÜ-HEM-HHT-02
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Nurse's Role; Mental Health Literacy; Education
Keywords: nursing educations; mental health literacy; creative drama

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: İn this study, the names of the patients nursing student in the two wards will be sorted and numbered in alphabetical order. After the numbering process, the patients will be selected to the experimental and control group by using the "www.randomizer.org/" site by an independent specialist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mental health literacy training supported by creative drama (Experimental): nursing students will be given two hours of mental health literacy training supported by creative drama one day a week for 4 weeks.
  Interventions: Other: mental health literacy training supported by creative drama
- mental health literacy training supported by classroom instruction (Experimental): nursing students will be given mental health literacy training supported by two hours of classroom instruction one day a week for 4 weeks.
  Interventions: Other: mental health literacy training supported by classroom instruction

INTERVENTIONS:
Other: mental health literacy training supported by creative drama — nursing students will be given two hours of mental health literacy training supported by creative drama one day a week for 4 weeks.
  Arms: mental health literacy training supported by creative drama
Other: mental health literacy training supported by classroom instruction — nursing students will be given mental health literacy training supported by two hours of classroom instruction one day a week for 4 weeks.
  Arms: mental health literacy training supported by classroom instruction

SUMMARY:
This study was planned as a randomized controlled trial to determine the effect of creative drama education given to nursing students on mental health literacy scores

DETAILED DESCRIPTION:
This studies designed experimentally. among the first-year students of nursing who cannot repeat the class, who have not received mental health literacy training before, and who are willing to participate in the study will form the group of the study. The designated group will be divided into experimental (creative drama) and control group (classroom training). Training to the experimental group will be applied to the control group through creative drama through in-f training. The trainings are planned as 4 sessions and each session/lesson is planned as 50+50 (100 minutes). As a measurement tool, the mental health literacy scale will be used as the pre-test and final test.

ELIGIBILITY:
Inclusion Criteria:

Have not received any training on mental health or mental health literacy, Have reached the age of 18 No more class repetition volunteer to participate in the study nursing students were included in the study

Exclusion Criteria:

Have received any training in mental health or mental health literacy, Under 18 years of age Remaining for class repetition who is not willing to participate in the study nursing students were not included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
experimental group (creative drama) nursing students' mental health literacy pretest final test scores | 21 Day
  Mental Health Literacy Scale (RSOS): The scale allows individuals to determine their RSO level and to determine in which areas they may need more support. The scale consists of sub-sub-dimensions of 35 items. The first 15 (1-15) items are quad likert (strongly disagree (1), disagree (2), agree (3), strongly agree (4)) and the next 20 (16-35) items are quintessentially likert (1), disagree (2), disagree (2), agree (3), agree (4), strongly agree (5).
Control group (classroom instruction) nursing students' mental health literacy pretest final test scores | 21 Day
  Mental Health Literacy Scale (RSOS): The scale allows individuals to determine their RSO level and to determine in which areas they may need more support. The scale consists of sub-sub-dimensions of 35 items. The first 15 (1-15) items are quad likert (strongly disagree (1), disagree (2), agree (3), strongly agree (4)) and the next 20 (16-35) items are quintessentially likert (1), disagree (2), disagree (2), agree (3), agree (4), strongly agree (5).

CONTACTS AND LOCATIONS:
Overall Officials: Hümeyra Hançer tok, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University- Faculty of Health Sciences- Department of Nursing, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study is planned as an individual research and will be presented as a publication in a journal.
Supporting Information: SAP
Time Frame: Data will be collected for 12 month
Access Criteria: you can contact the author

REFERENCES:
- [Result] Faigenbaum AD, Rebullido TR, Zaichkowsky L. Heads-up: Effective Strategies for Promoting Mental Health Literacy in Youth Fitness Programs. ACSMs Health Fit J. 2022;26(3):12-9.
- [Result] Akgun S, Kesgin MT, Tok HH, Uzun LN. Comparison of Psychological Distress and Mental Health Literacy Levels of Hospitalized COVID-19 Patients, Individuals under Quarantine, and Healthy Individuals of Society in The Pandemic. ASEAN Journal of Psychiatry. 2021;22(8):1-11.
- [Result] Milin R, Kutcher S, Lewis SP, Walker S, Wei Y, Ferrill N, Armstrong MA. Impact of a Mental Health Curriculum on Knowledge and Stigma Among High School Students: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 May;55(5):383-391.e1. doi: 10.1016/j.jaac.2016.02.018. Epub 2016 Mar 8. PMID 27126852
- [Result] Özoğul T, Sezerel H, Aktaş SG, Adıgüzel Ö. Learning through creative drama in vocational hospitality education: Efficiency, retention, and attitudes. Tour Manag Perspect. 2020;36:100728.